CLINICAL TRIAL: NCT05511870
Title: A Single Center, Randomized, Double-Blind, Placebo-Controlled Phase 1 Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Etripamil in Healthy Chinese Subjects
Brief Title: A Study of Etripamil in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: JX02001
Record Dates: First submitted 2022-08-07; First posted 2022-08-23 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Healthy Chinese Subjects
Keywords: Etripamil; Paroxysmal supraventricular tachycardia; Tachycardia; Tachycardia, Supraventricular
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia; Tachycardia, Supraventricular

STUDY DESIGN:
Intervention Model Description: A Single Center, Randomized, Double-Blind, Placebo-Controlled Phase 1 Study
Who Masked: Participant, Investigator
Masking Description: JX02001 is a double blind phase 1 study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etripamil Nasal Spray 70mg (Experimental): Etripamil Nasal Spray 70mg single dose
  Interventions: Drug: Etripamil Nasal Spray 70mg
- Etripamil Placebo Nasal Spray 70mg (Placebo Comparator): Etripamil Placebo Nasal Spray 70mg single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etripamil Nasal Spray 70mg — Etripamil NS 70 mg will be administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Arms: Etripamil Nasal Spray 70mg
Drug: Placebo — Placebo will be administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Arms: Etripamil Placebo Nasal Spray 70mg

SUMMARY:
The objectives of the study are as below:

Primary:

·To evaluate the pharmacokinetics (PK) of Etripamil in healthy adult Chinese subjects

Secondary:

* To evaluate the pharmacodynamics (PD) of Etripamil in healthy adult Chinese subjects
* To evaluate the safety and tolerability of Etripamil in healthy adult Chinese subjects

Exploratory:

·To evaluate the PK exposure-PD response relationship of etripamil in healthy adult Chinese subjects

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase 1 study in healthy adult Chinese subjects to evaluate the PK, PD, safety and tolerability of single dose of etripamil, 70 mg nasal spray (NS). After signing the informed consent form (ICF), potential subjects will undergo screening procedures within 28 days prior to dosing. Eligible subjects will be admitted to the clinical unit on Day -1 and screening procedures will be repeated to confirm eligibility. Subjects will fast overnight for at least 10 hours prior to dosing. 12 healthy adult Chinese subjects will be randomized to receive etripamil 70 mg single dose (n=10) or placebo (n=2).

Blood and urine samples will be collected for PK assessments of etripamil and the inactive main metabolite MSP-2030.

AEs, 12-lead ECGs, clinical laboratory tests, vital signs, physical examinations, and concomitant medications will be collected and evaluated over the course of study.

Subjects will remain in clinic until discharged on Day 2. There will be a follow-up telephone call on Day 11 (±1 day) of dosing. Total duration for each subject will be approximately 1.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all the following criteria at screening may be included in the study:

  1. Ethnically Chinese men or women, 18 to 45 years of age (inclusive).
  2. Body weight: male ≥50 kg, female ≥45 kg; body mass index (BMI) within 18 to 26 kg/m2 (inclusive).
  3. Healthy subject as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital signs.
  4. Able to comprehend and willing to sign the ICF which includes compliance with the inclusion and exclusion criteria listed in the ICF and in the protocol.
  5. Non-smoker or ex-smoker for >6 months.
  6. From the time they sign the informed consent to 90 days (male subject within 30 days) after dosing, subjects have no plans to have children and voluntarily use effective contraception

Exclusion Criteria:

* Any of the following will exclude subjects from the study:

  1. Have a history of, or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal disease; thyroid disease; neurologic or psychiatric disease; or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results.
  2. A history of atrioventricular (AV) block, (1st, 2nd or 3rd degree), myocardial infarction (MI) or angina, non-sustained or sustained ventricular tachycardia (VT), torsade de pointes, family history of sudden death or prolonged QT interval, vaso-vagal syncope, sick sinus syndrome, supraventricular tachycardia, atrial flutter, atrial fibrillation (AFib), stroke, transient ischemic attack (TIA), unexplained syncope, congestive heart failure (CHF).
  3. Acute upper respiratory tract infection within 14 days prior to dosing.
  4. Any abnormality of the nasal passage.
  5. Unable to tolerate IN administration.
  6. Known sensitivity to verapamil or other drugs or foods.
  7. Clinically significant abnormal values for clinical laboratory tests at screening as deemed appropriate by the investigator.
  8. Serum potassium <3.5mmol/L or serum magnesium <0.75mmol/L or serum calcium <2.11mmol/L.
  9. Systolic blood pressure (SBP) <100 or >140 mmHg, diastolic blood pressure (DBP) <55 or >90 mmHg, HR <65 or >95 bpm.
  10. QTcF >440 msec, flat or biphasic T waves, QRS >105 ms, evidence of a prior MI, pathologic U waves or U waves that interfere with the QT measurement, AV block or left anterior hemiblock (LAHB) or left posterior hemiblock (LPHB) or right bundle branch block (RBBB) or left bundle branch block (LBBB), pre-excitation syndrome.
  11. Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening as deemed appropriate by the Investigator.
  12. Have a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; have a history of treponema pallidum antibody positive, or tests positive for treponema pallidum; have a history of hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCVAb) positive, or other clinically active liver disease, or tested positive for HBsAg or HCVAb at screening.
  13. History of drug or alcohol abuse in the last 2 years..
  14. Positive test result(s) for alcohol and/or drugs of abuse at screening or admission (Day-1).
  15. Received an investigational drug or used an invasive investigational medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before dosing.
  16. Use of any prescription or non-prescription medication within 14 days or 5 half-lives (whichever is longer), or complementary and alternative medicine within 28 days before dosing (excluding aspirin, ibuprofen, and acetaminophen).
  17. Any blood donation within 60 days prior to dosing, or any plasma donation within 30 days prior to dosing, or receipt of blood products within 60 days prior to dosing.
  18. Vaccinated within 30 days prior to dosing or planned to be vaccinated during this study.
  19. Have preplanned surgery or procedures that will interfere with the conduct of the study.
  20. Sponsor staff and/or staff at the study site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Cmax of Etripamil after single dosing | Day -1 to Day 11
  To measure Cmax of Etripamil after single dosing
Cmax of MSP-2030 after single dosing | Day -1 to Day 11
  To measure Cmax of MSP-2030 after single dosing

SECONDARY OUTCOMES:
PR interval after single dosing | Day -1 to Day 11
  To measure PR interval by electrocardiogram after single dosing
Blood pressure after single dosing | Day -1 to Day 11
  To measure systolic and diastolic blood pressure after single dosing
Heart rate after single dosing | Day -1 to Day 11
  To measure heart rate after single dosing
Subject incidence of Adverse Event (AE) | Day -1 to Day 11
  To record subject incidence of Adverse Event (AE)
Subject electrocardiogram outcomes | Day -1 to Day 11
  To record number of participants with abnormal electrocardiogram readings
Subject clinical laboratory tests outcomes | Day -1 to Day 11
  To record number of participants with abnormal laboratory test results
Concomitant medications that subjects take | Day -1 to Day 11
  To record subject clinical laboratory tests outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jing ZHANG, Principal Investigator — Huashan Hospital; Yuewen XI, Principal Investigator — Huashan Hospital; Lihang QI, Study Director — Corxel Pharmaceuticals
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China